CLINICAL TRIAL: NCT04529837
Title: Longitudinal Ultrasound Evaluation of Dilapan-S During Cervical Ripening
Brief Title: Ultrasound Assessment of DILAPAN-S
Status: Completed | Type: Observational
Sponsor: Eastern Virginia Medical School (Other)
Responsible Party: Principal Investigator, Elizabeth Seagraves, Maternal Fetal Medicine Fellow, Eastern Virginia Medical School
Other Study IDs: 20-40-FB-0097
Record Dates: First submitted 2020-08-17; First posted 2020-08-28 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Cervical Dilation; Induction of Labor; Ultrasound Evaluation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Pregnant individuals with Dilapan-S only: 22 women received Dilapan-S rods without gauze at start of induction.
  Interventions: Other: No gauze
- Pregnant individuals with Dilapan-S plus gauze placement: 22 women received Dilapan-S rods with 1 gauze at start of induction.
  Interventions: Other: Gauze

INTERVENTIONS:
Other: Gauze — placement of gauze
  Groups: Pregnant individuals with Dilapan-S plus gauze placement
Other: No gauze — no gauze
  Groups: Pregnant individuals with Dilapan-S only

SUMMARY:
The goal of this observational prospective study is to assess the change in Dilapan-S rod diameters using transvaginal ultrasound over a period of 12 hours in term women undergoing induction of labor.

DETAILED DESCRIPTION:
On admission for induction, study participants assigned to each group underwent continuous cardiotocography for 20 minutes prior to placement of the Dilapan-S rods (rod size: 4 x 65mm). Placement of the Dilapan-S rods was limited to three physicians with the majority placed by the primary investigator. Placement was completed in a sterile manner under direct visualization and in accordance with the manufacturer's guidelines. The number of rods placed varied per individual and was based on the discretion of the physician. Each participant allocated to the Dilapan-S with saturated gauze group received placement of one, 4x4 inch gauze saturated with 10 cc of normal saline and placed at the level of the external os. Immediately after placement of the Dilapan-S rods, the study participant was asked to complete a patient satisfaction survey.

Pre-specified transvaginal ultrasound assessment was performed at hours 3, 6, 8, and 12 post Dilapan-S placement using a GE Voluson E10 machine with a transvaginal GE RIC 5-9D transducer. Performance of the ultrasound evaluation was limited to the primary investigator and two co-authors of the study. After completion of the 12-hour ultrasound, the Dilapan-S rods and gauze, if used, were removed as per the manufacturer's instructions. The participant was then asked to complete a post Dilapan-S patient satisfaction survey.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant individuals at gestational age 37 weeks or greater.
* Scheduled medical or elective induction at Sentara Norfolk General Hospital.
* Live, singleton IUP.
* Vertex presentation.
* Intact membranes.
* Bishop score of 6 or less.

Exclusion Criteria:

* Unwilling or unable to provide consent.
* Intrauterine fetal demise
* Contraindications to vaginal delivery.
* BMI > 45
* Vaginal bleeding
* Clinically evident genital tract infection

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant individuals at term undergoing labor induction at single academic institution.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Diameter change of Dilapan-S | 12 hours
  Rod diameters of Dilapan-S rods were measured via transvaginal ultrasound at 3,6,8, and 12 hours after placement.

SECONDARY OUTCOMES:
Gauze placement and rod diameter | 12 hours
  Rod diameters of Dilapan-S rods plus gauze placement were measured via transvaginal ultrasound at 3,6,8, and 12 hours after placement.
Patient satisfaction | 12 hours
  Patient satisfaction scores were assessed based on gauze versus no gauze placement.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Seagraves, DO, Principal Investigator — Eastern Virginia Medical School MFM Fellowship
Locations (1):
- Eastern Virginia Medical School, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, statistical analysis plan, informed consent form were made available. Results from the study will be available to the manufacturer (Medicem) after statistical analysis is completed and will not be shared with the manufacturer during study execution. The manufacturer company will not be involved in data analysis and all data will be independently analyzed by HADSI. The results of this study will be presented at conferences or published in a peer-review journal.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1-2 months after conclusion of study
Access Criteria: Results and statistical analysis will be available at the conclusion of the study

REFERENCES:
- [Background] Chen W, Xue J, Peprah MK, Wen SW, Walker M, Gao Y, Tang Y. A systematic review and network meta-analysis comparing the use of Foley catheters, misoprostol, and dinoprostone for cervical ripening in the induction of labour. BJOG. 2016 Feb;123(3):346-54. doi: 10.1111/1471-0528.13456. Epub 2015 Nov 5. PMID 26538408
- [Background] Grobman WA, Rice MM, Reddy UM, Tita ATN, Silver RM, Mallett G, Hill K, Thom EA, El-Sayed YY, Perez-Delboy A, Rouse DJ, Saade GR, Boggess KA, Chauhan SP, Iams JD, Chien EK, Casey BM, Gibbs RS, Srinivas SK, Swamy GK, Simhan HN, Macones GA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Labor Induction versus Expectant Management in Low-Risk Nulliparous Women. N Engl J Med. 2018 Aug 9;379(6):513-523. doi: 10.1056/NEJMoa1800566. PMID 30089070
- [Background] American College of Obstetricians and Gynecologists. Induction of Labor. ACOG Practice Bulletin No. 107. August 2009.
- [Background] Saad AF, Villarreal J, Eid J, Spencer N, Ellis V, Hankins GD, Saade GR. A randomized controlled trial of Dilapan-S vs Foley balloon for preinduction cervical ripening (DILAFOL trial). Am J Obstet Gynecol. 2019 Mar;220(3):275.e1-275.e9. doi: 10.1016/j.ajog.2019.01.008. Epub 2019 Feb 18. PMID 30790569
- [Background] Drunecky T, Reidingerova M, Plisova M, Dudic M, Gdovinova D, Stoy V. Experimental comparison of properties of natural and synthetic osmotic dilators. Arch Gynecol Obstet. 2015 Aug;292(2):349-54. doi: 10.1007/s00404-015-3623-3. Epub 2015 Jan 25. PMID 25618749
- [Background] Gupta J, Chodankar R, Baev O, Bahlmann F, Brega E, Gala A, Hellmeyer L, Hruban L, Maier J, Mehta P, Murthy A, Ritter M, Saad A, Shmakov R, Suneja A, Zahumensky J, Gdovinova D. Synthetic osmotic dilators in the induction of labour-An international multicentre observational study. Eur J Obstet Gynecol Reprod Biol. 2018 Oct;229:70-75. doi: 10.1016/j.ejogrb.2018.08.004. Epub 2018 Aug 3. PMID 30107363
- [Background] Chambers DG, Willcourt RJ, Laver AR, Baird JK, Herbert WY. Comparison of Dilapan-S and laminaria for cervical priming before surgical pregnancy termination at 17-22 weeks' gestation. Int J Womens Health. 2011;3:347-52. doi: 10.2147/IJWH.S25551. Epub 2011 Oct 20. PMID 22114527
- [Background] Abuhamad, A. Ultrasound in Obstetrics and Gynecology: A Practical Approach. Chapter 1: Basic Physical Principles of Medical Ultrasound. 2014.
- [Background] Sung YT, Wu JS. The Visual Analogue Scale for Rating, Ranking and Paired-Comparison (VAS-RRP): A new technique for psychological measurement. Behav Res Methods. 2018 Aug;50(4):1694-1715. doi: 10.3758/s13428-018-1041-8. PMID 29667082
- [Background] Kliger M, Stahl S, Haddad M, Suzan E, Adler R, Eisenberg E. Measuring the Intensity of Chronic Pain: Are the Visual Analogue Scale and the Verbal Rating Scale Interchangeable? Pain Pract. 2015 Jul;15(6):538-47. doi: 10.1111/papr.12216. Epub 2014 Apr 16. PMID 24735056
- See also: Recent declines in induction of labor by gestational age — https://www.cdc.gov/nchs/products/databriefs/db155.htm.
- See also: Women's Health Fastfacts — https://www.cdc.gov/nchs/fastats/womens-health.htm